CLINICAL TRIAL: NCT03987139
Title: Cerebral Autoregulation in Patients With Aneurysmal SubArachnoid Haemorrhage
Acronym: CASAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Markus Harboe Olsen, Research Fellow, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: H-19017185
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
Keywords: cerebral autoregulation
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Intervention is performed once in both patients (after the aneurysm is closed and max. 5 days after ictus) and controls. The procedure consists of the following sessions:
  1. Induced hypertension; as well
  2. (Only in mechanically ventilated patients) either
     1. Mild hyper- and hypocapnia or
     2. Mild hyper- and hypoxia.
  In session 2 (hyper- / hypoxia or hyper- / hypocapnia), patients are randomized to order the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): Patients included in the study.
  Interventions: Other: Hypertension; Other: Hyper- and hypoxia; Other: Hyper- and hypocapnia

INTERVENTIONS:
Other: Hypertension — Hypertension is induced by an infusion of noradrenaline within acceptable limits Baseline recording (10 minutes) is performed. MAP gradually increases in steps of 5-10 mmHg during ongoing TCD. When the desired maximum MAP is reached, measurement is made at steady state (10 minutes).
  Noradrenaline infusion is stopped. When MAP is stabilized, new baseline is measured for 10 minutes.
Other: Hyper- and hypoxia — The mechanical ventilator is adjusted to mild hypoxia, normoxia and mild hyperoxia. Measurements are made for 10 minutes at normoxia and after steady state is reached, respectively. hyperoxia and hypoxia. Oxygenation is controlled by arterial blood gas before and during steady state.
Other: Hyper- and hypocapnia — The mechanical ventilator is adjusted to a delta PaCO2 on the ventilator for both hypocapnia and hypercapnia. Measurements are made for 10 minutes at normocapnia and after steady state is reached, respectively. hyper- and hypocapnia.

SUMMARY:
The purpose is, in patients with aneurysmal subarachnoid haemorrhage in the early phase after ictus, to examine the following:

1. The effect of spontaneous and induced changes on the brain's static and dynamic autoregulation calculated by transcranial Doppler (TCD), ICP and MAP (primary purposes) and ICP and PbtO2;
2. The effect of mild hyper- and hypocapnia as well as of mild hyper- and hypoxia on the brain's static and dynamic autoregulation, ICP and PbtO2;
3. The relationship between brain autoregulation, mild hyper- and hypocapnia, as well as of mild hyper- and hypoxia and metabolism in microdialysate on the one hand and the occurrence of DCI during hospitalization and poor neurological outcome one year after ictus on the other.

DETAILED DESCRIPTION:
Spontaneous aneurysm subarachnoid hemorrhage (SAH) occurs annually in approximately 400 people in Denmark. SAH is most commonly seen in younger (median age 56 years) and women (71%), have a high mortality (21-44%) and result in a poor neurological outcome in about 50% of patients. Due to the relatively young patient population and high mortality and morbidity, SAH in the population causes the same number of lost working years as blood clots in the brain.

The occurrence of complications like hydrocephalus and re-bleeding can be minimized by rapid external ventricular drainage and aneurysm closure, and so-called delayed cerebral ischaemia (DCI) is currently considered to be the most frequent serious complication of SAH. DCI occurs in 20-30% of patients, most often within the first 14 days, is characterized by a reduction in consciousness or focal neurological deficit lasting at least one hour without any other underlying cause and is associated with a significantly increased risk of a poor outcome. The cause and treatment of DCI is controversial, and the previous hypothesis of vasospasm as the sole contributor is currently supplemented by a broader focus on several other mechanisms, including the brain's blood supply and its regulation.

The brain's blood supply (CBF) is kept relatively constant in healthy by changing cardiac diameter and thus the cerebrovascular resistance (CVR) during changes in brain perfusion pressure (CPP, measured as mean arterial pressure (MAP) minus intracranial pressure (ICP)) within certain limits. This mechanism is known as cerebral autoregulation. Outside these limits, respectively. decreases and increases CBF, with the consequent risk of hypoperfusion/ischemia and hyperperfusion/vasogenic edema with prolonged changes.

Weakened autoregulation, i.e. that CBF varies passively with CPP also within the normal autoregulation limits, is described in e.g. traumatic brain injury (TBI), ischemic stroke, acute liver failure and meningitis, with complete or partial restoration of autoregulation by hyperventilation (mild hypocapnia). SAH also describes impaired autoregulation with varying association with disease severity, DCI and outcome. It is not known whether mild hypocapnia restores autoregulation in patients with SAH, whereas animal experimental studies suggest this.

Reduced intracerebral oxygenation (PbtO2) is associated with a worse outcome after SAH. Cerebral microdialysis measures the concentration of certain metabolites in the brain and can provide an insight into whether metabolic activity is affected by oxygen deficiency, and so-called anaerobic combustion occurs. Microdialysis measurements with elevated lactate concentration, which is a metabolic product, among other things. Anaerobic combustion appears to occur prior to clinical signs of DCI, as well as during the DCI episodes, decreasing PbtO2. It is possible that these findings could be due to a condition of impaired autoregulation and too low perfusion pressure to meet brain metabolic needs, but this has not previously been elucidated. It is also unknown if it is possible to improve brain metabolism by increasing the brain's perfusion pressure.

The purpose of this study is therefore to investigate brain autoregulation in patients with SAH.

ELIGIBILITY:
Inclusion Criteria, patients:

* Admittance to neurointensive care unit, Rigshospitalet
* Age ≥ 18 years old
* Aneurysmal subarachnoid haemorrhage
* Clinical indication for placement of an external ventricular drain
* Measurements can be done within 3 days of ictus
* Closest relatives understand written and spoken danish

Exclusion Criteria, patients:

* No aneurysm identified
* Conservative og failed treatment of aneurysm
* Pupils dilated and do not react to light
* Incarceration before inclusion
* Expected death within 48 hours
* Acute or chronic diseases associated with impaired autoregulation
* Severe chronic lung failure with a PaCO2 > 6.5 kPa or PaO2 < 8 kPa.

Inclusion Criteria, healthy subjects:

* Age ≥ 18 years old;
* Understands written and spoken danish
* Oral and written consent
* No medication expect hay fever medications
* Alcohol consumption within the limits from the danish health care board
* Healthy without previous or current cerebrovascular diseases
* Insonation is possible from the middle cerebral artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Middle cerebral artery flow velocity (MCAv) + induced hypertension | within 5 days after ictus, for 10 minutes after steady state
  Measuring MCAv after induced hypertension

SECONDARY OUTCOMES:
Intracranial pressure (ICP) + induced hypertension | within 5 days after ictus
  Measuring changes in ICP after induced hypertension
Partial brain tissue oxygenation (PbtO2) + induced hypertension | within 5 days after ictus
  Measuring changes in ICP after induced hypertension
Intracranial pressure (ICP) + hyper- and hypocapnia | within 5 days after ictus, for 10 minutes after steady state
  Measuring during induction of hyper- and hypocapnia
Partial brain tissue oxygenation (PbtO2) + hyper- and hypocapnia | within 5 days after ictus, for 10 minutes after steady state
  Measuring during induction of hyper- and hypocapnia
Intracranial pressure (ICP) + hyper- and hypoxia | within 5 days after ictus, for 10 minutes after steady state
  Measuring during induction of hyper- and hypoxia
Partial brain tissue oxygenation (PbtO2) + hyper- and hypoxia | within 5 days after ictus, for 10 minutes after steady state
  Measuring during induction of hyper- and hypoxia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroanaesthesiology, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data from each individual participant will be available after publication of planned manuscripts, with a valid reason, and after signing a data processing agreement.
Supporting Information: Study Protocol
Time Frame: The approved study protocol will be available upon request until publication of the study results
Access Criteria: Valid reason and contact with author

REFERENCES:
- [Background] Kurian MA, Li Y, Zhen J, Meyer E, Hai N, Christen HJ, Hoffmann GF, Jardine P, von Moers A, Mordekar SR, O'Callaghan F, Wassmer E, Wraige E, Dietrich C, Lewis T, Hyland K, Heales S Jr, Sanger T, Gissen P, Assmann BE, Reith ME, Maher ER. Clinical and molecular characterisation of hereditary dopamine transporter deficiency syndrome: an observational cohort and experimental study. Lancet Neurol. 2011 Jan;10(1):54-62. doi: 10.1016/S1474-4422(10)70269-6. Epub 2010 Nov 25. PMID 21112253
- [Background] Olsen MH, Orre M, Leisner ACW, Rasmussen R, Bache S, Welling KL, Eskesen V, Moller K. Delayed cerebral ischaemia in patients with aneurysmal subarachnoid haemorrhage: Functional outcome and long-term mortality. Acta Anaesthesiol Scand. 2019 Oct;63(9):1191-1199. doi: 10.1111/aas.13412. Epub 2019 Jun 7. PMID 31173342
- [Background] van Gijn J, Kerr RS, Rinkel GJ. Subarachnoid haemorrhage. Lancet. 2007 Jan 27;369(9558):306-18. doi: 10.1016/S0140-6736(07)60153-6. PMID 17258671
- [Background] Brathwaite S, Macdonald RL. Current management of delayed cerebral ischemia: update from results of recent clinical trials. Transl Stroke Res. 2014 Apr;5(2):207-26. doi: 10.1007/s12975-013-0316-8. Epub 2013 Dec 13. PMID 24338266
- [Background] Schmidt JM, Wartenberg KE, Fernandez A, Claassen J, Rincon F, Ostapkovich ND, Badjatia N, Parra A, Connolly ES, Mayer SA. Frequency and clinical impact of asymptomatic cerebral infarction due to vasospasm after subarachnoid hemorrhage. J Neurosurg. 2008 Dec;109(6):1052-9. doi: 10.3171/JNS.2008.109.12.1052. PMID 19035719
- [Background] Dankbaar JW, Slooter AJ, Rinkel GJ, Schaaf IC. Effect of different components of triple-H therapy on cerebral perfusion in patients with aneurysmal subarachnoid haemorrhage: a systematic review. Crit Care. 2010;14(1):R23. doi: 10.1186/cc8886. Epub 2010 Feb 22. PMID 20175912
- [Background] Roos YB, de Haan RJ, Beenen LF, Groen RJ, Albrecht KW, Vermeulen M. Complications and outcome in patients with aneurysmal subarachnoid haemorrhage: a prospective hospital based cohort study in the Netherlands. J Neurol Neurosurg Psychiatry. 2000 Mar;68(3):337-41. doi: 10.1136/jnnp.68.3.337. PMID 10675216
- [Background] Dorhout Mees SM, Kerr RS, Rinkel GJ, Algra A, Molyneux AJ. Occurrence and impact of delayed cerebral ischemia after coiling and after clipping in the International Subarachnoid Aneurysm Trial (ISAT). J Neurol. 2012 Apr;259(4):679-83. doi: 10.1007/s00415-011-6243-2. Epub 2011 Sep 24. PMID 21947244
- [Background] Budohoski KP, Czosnyka M, Kirkpatrick PJ, Smielewski P, Steiner LA, Pickard JD. Clinical relevance of cerebral autoregulation following subarachnoid haemorrhage. Nat Rev Neurol. 2013 Mar;9(3):152-63. doi: 10.1038/nrneurol.2013.11. Epub 2013 Feb 19. PMID 23419369
- [Background] Macdonald RL. Delayed neurological deterioration after subarachnoid haemorrhage. Nat Rev Neurol. 2014 Jan;10(1):44-58. doi: 10.1038/nrneurol.2013.246. Epub 2013 Dec 10. PMID 24323051
- [Background] LASSEN NA. Cerebral blood flow and oxygen consumption in man. Physiol Rev. 1959 Apr;39(2):183-238. doi: 10.1152/physrev.1959.39.2.183. No abstract available. PMID 13645234
- [Background] Berg, R.M.G., Pedersen, M., Møller, K.: Static cerebral blood flow autoregulation in humans. Curr. Hypertens. Rev. 5, 140-157 (2009).
- [Background] Czosnyka M, Smielewski P, Piechnik S, Steiner LA, Pickard JD. Cerebral autoregulation following head injury. J Neurosurg. 2001 Nov;95(5):756-63. doi: 10.3171/jns.2001.95.5.0756. PMID 11702864
- [Background] Eames PJ, Blake MJ, Dawson SL, Panerai RB, Potter JF. Dynamic cerebral autoregulation and beat to beat blood pressure control are impaired in acute ischaemic stroke. J Neurol Neurosurg Psychiatry. 2002 Apr;72(4):467-72. doi: 10.1136/jnnp.72.4.467. PMID 11909905
- [Background] Strauss G, Hansen BA, Knudsen GM, Larsen FS. Hyperventilation restores cerebral blood flow autoregulation in patients with acute liver failure. J Hepatol. 1998 Feb;28(2):199-203. doi: 10.1016/0168-8278(88)80006-0. PMID 9514532
- [Background] Moller K, Skinhoj P, Knudsen GM, Larsen FS. Effect of short-term hyperventilation on cerebral blood flow autoregulation in patients with acute bacterial meningitis. Stroke. 2000 May;31(5):1116-22. doi: 10.1161/01.str.31.5.1116. PMID 10797174
- [Background] Otite F, Mink S, Tan CO, Puri A, Zamani AA, Mehregan A, Chou S, Orzell S, Purkayastha S, Du R, Sorond FA. Impaired cerebral autoregulation is associated with vasospasm and delayed cerebral ischemia in subarachnoid hemorrhage. Stroke. 2014 Mar;45(3):677-82. doi: 10.1161/STROKEAHA.113.002630. Epub 2014 Jan 14. PMID 24425120
- [Background] Budohoski KP, Czosnyka M, Kirkpatrick PJ, Reinhard M, Varsos GV, Kasprowicz M, Zabek M, Pickard JD, Smielewski P. Bilateral failure of cerebral autoregulation is related to unfavorable outcome after subarachnoid hemorrhage. Neurocrit Care. 2015 Feb;22(1):65-73. doi: 10.1007/s12028-014-0032-6. PMID 25056137
- [Background] Ma X, Willumsen L, Hauerberg J, Pedersen DB, Juhler M. Effects of graded hyperventilation on cerebral blood flow autoregulation in experimental subarachnoid hemorrhage. J Cereb Blood Flow Metab. 2000 Apr;20(4):718-25. doi: 10.1097/00004647-200004000-00009. PMID 10779016
- [Background] Ramakrishna R, Stiefel M, Udoetuk J, Spiotta A, Levine JM, Kofke WA, Zager E, Yang W, Leroux P. Brain oxygen tension and outcome in patients with aneurysmal subarachnoid hemorrhage. J Neurosurg. 2008 Dec;109(6):1075-82. doi: 10.3171/JNS.2008.109.12.1075. PMID 19035722
- [Background] Skjoth-Rasmussen J, Schulz M, Kristensen SR, Bjerre P. Delayed neurological deficits detected by an ischemic pattern in the extracellular cerebral metabolites in patients with aneurysmal subarachnoid hemorrhage. J Neurosurg. 2004 Jan;100(1):8-15. doi: 10.3171/jns.2004.100.1.0008. PMID 14743906
- [Background] Roh DJ, Morris NA, Claassen J. Intracranial Multimodality Monitoring for Delayed Cerebral Ischemia. J Clin Neurophysiol. 2016 Jun;33(3):241-9. doi: 10.1097/WNP.0000000000000277. PMID 27258448
- [Derived] Olsen MH, Capion T, Riberholt CG, Bache S, Ebdrup SR, Rasmussen R, Mathiesen T, Berg RMG, Moller K. Effect of controlled blood pressure increase on cerebral blood flow velocity and oxygenation in patients with subarachnoid haemorrhage. Acta Anaesthesiol Scand. 2023 Sep;67(8):1054-1060. doi: 10.1111/aas.14277. Epub 2023 May 16. PMID 37192754